CLINICAL TRIAL: NCT01554085
Title: A Randomized, Double-blind, Placebo-controlled, First-in-human, 3-Part Study of Orally Administered ALS-002158 to Evaluate the Safety, Tolerability and Pharmacokinetics of Single Ascending Dosing and Food-effect in Healthy Volunteers, and Multiple Ascending Dosing in Subjects With Chronic Hepatitis C Genotype 1 Infection
Brief Title: First in Human Study of ALS-002158; Single Dose, Food Effect in Healthy Volunteers; Multiple Doses in Chronic Hepatitis C Genotype 1
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: ALS-2158 showed insufficient antiviral activity to warrant proceeding with further clinical development.
Sponsor: Alios Biopharma Inc. (Industry)
Collaborators: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALS-2158-201
Record Dates: First submitted 2012-03-12; First posted 2012-03-14 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

ARMS (2):
- ALS-002158 (Experimental)
  Interventions: Drug: ALS-002158
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALS-002158 — ALS-002158
  Arms: ALS-002158
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, 3-part study will assess the safety, tolerability, and pharmacokinetics of orally administered ALS-002158 in healthy volunteers (HV) and subjects with chronic hepatitis C (CHC) genotype 1 infection.

Part 1 will assess single ascending dosing pharmacokinetics and safety in HV. Part 2 will assess food effects on pharmacokinetics in HV.

Part 3 will assess multiple ascending dosing pharmacokinetics and safety in subjects with CHC genotype 1 infection.

ELIGIBILITY:
Inclusion Criteria:

* Subject has provided written consent.
* Subject is in good health as deemed by the investigator
* Creatinine clearance of greater than 50 mL/min (Cockcroft- Gault).
* Male or female, 18-55 years of age for HV and 18-65 years of age for subjects with CHC.
* Body mass index (BMI) 18-32 kg/m2 inclusive for HV and 18-36 kg/m2 for subjects with CHC, minimum weight 50 kg in both populations.
* A female is eligible to participate in this study if she is of non-childbearing potential.
* If male, subject is surgically sterile or practicing specific forms of birth control.

Additional inclusion criteria for subjects with CHC genotype 1 infection:

* Positive HCV antibody and a positive HCV RNA at screening.
* Documentation of CHC infection of greater than 6 months duration at screening.
* CHC genotype 1 infection at screening.
* HCV RNA viral load ≥ 105 and ≤ 108 IU/mL using a sensitive quantitative assay
* Liver biopsy within two years or Fibroscan evaluation within 6 months prior to screening that clearly excludes cirrhosis. Fibroscan liver stiffness score must be < 12 kPa.
* Absence of hepatocellular carcinoma as indicated by an abdominal ultrasound scan during screening.
* No prior treatment for CHC.
* Absence of history of clinical hepatic decompensation.
* Laboratory values include:

  * prothrombin time < 1.5 × ULN.
  * platelets > 120,000/mm3.
  * albumin > 3.5 g/dL, bilirubin < 1.5 mg/dL at screening (subjects with documented Gilbert's disease allowed).
  * Serum ALT concentration < 5 × ULN.
  * Alpha Fetoprotein (AFP) concentration ≤ ULN. If AFP is ≥ ULN, absence of a hepatic mass must be demonstrated by ultrasound within the screening period.

Exclusion Criteria:

* Clinically significant cardiovascular, respiratory, renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder.
* Positive test for HAV IgM, HBsAg, HCV Ab (HV only), or HIV Ab.
* Abnormal screening laboratory results that are considered clinically significant by the investigator.
* Clinically significant drug allergy such as, but not limited to, sulfonamides and penicillins, including those experienced in previous trials with experimental drugs.
* Participation in an investigational drug trial or having received an investigational vaccine within 30 days or 5 half lives (whichever is longer) prior to receiving study medication.
* Clinically significant blood loss or elective blood donation of significant volume.
* Laboratory abnormalities including:

  * Thyroid Stimulating Hormone (TSH) >ULN.
  * Hematocrit < 34 %.
  * White blood cell counts < 3,500/mm3.
* For healthy volunteers, history of regular use of tobacco.
* The subject has a positive pre-study drug screen.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2011-12-31 (Actual); Primary Completion 2012-09-30 (Actual); Study Completion 2012-09-30 (Actual)

PRIMARY OUTCOMES:
Tabulation of adverse events, physical exam, vital signs, 12-lead ECGs, and clinical lab results | Part 1: Day 1-8; Part 2: Day 1-16; Part 3: Day 1-31

SECONDARY OUTCOMES:
Pharmacokinetic parameters and urinary excretion of ALS-002158 and metabolites | Part 1: Day 1-8; Part 2: Day 1-16; Part 3: Day 1-31
  Maximum measured drug concentration (Cmax), time of maximum concentration (tmax), half-life (t1/2), apparent oral clearance (CL/F), area under the concentration time curve from time zero to infinity (AUC0-inf) or area under the concentration time curve from time zero to last quantifiable concentration (AUC0-last), area under the concentration time curve during the dosing interval (AUC0-tau)
HCV ribonucleic acid (RNA) viral load reduction | Baseline to Day 31
Sequence analysis of the Hepatitis C virus (HCV) NS5B region | Baseline up to Month 6

CONTACTS AND LOCATIONS:
Locations (5):
- Australia (3):
  - QPharm, Brisbane, Queensland
  - CMAX, Adelaide, South Australia
  - Linear Clinical Research Ltd, Perth, Western Australia
- New Zealand (2):
  - Auckland Clinical Services, Auckland
  - Christchurch Clinical Studies Trust Ltd., Christchurch